CLINICAL TRIAL: NCT00005761
Title: Study of Association of Serum Factors With Diabetic Retinopathy
Brief Title: Blood Factors and Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000135; 00-EI-0135
Record Dates: First submitted 2000-05-26; First posted 2000-05-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-12-07

CONDITIONS: Diabetic Retinopathy
Keywords: Types 1 & 2 Diabetes; Cell Adhesion Molecules; Chemokines; Vascular Endothelial Growth Factor; Cross-Sectional; Serum Levels; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

SUMMARY:
This study will determine whether certain factors in the blood are associated with the severity of diabetic retinopathy.

Patients age 10 years and older with diabetes mellitus and diabetic retinopathy may be eligible for this study. Those enrolled will represent a range of diabetic retinopathy from minimal to severe. Participants will undergo the following procedures:

* medical history
* thorough eye examination
* photographs of the eye
* blood tests to measure blood lipids (cholesterol and triglycerides) and serum creatinine (for kidney function)
* blood tests to measure levels of blood factors (cell adhesion molecules, chemokines and vascular endothelial growth factor) that may be related to the progression of diabetic retinopathy
* blood pressure measurement
* urinalysis

This study may lead to a better understanding of how diabetic retinopathy develops and progresses.

DETAILED DESCRIPTION:
Participants with a range of severity of diabetic retinopathy and healthy volunteers will be evaluated once for serum levels of cell adhesion molecules, chemokines and vascular endothelial growth factor. This study may lead to a better understanding of the pathogenesis of diabetic retinopathy and the identifying of possible targets for treatment. All study participants will undergo an ocular exam and ophthalmic photography. Blood is drawn for the analysis of these serum factors.

ELIGIBILITY:
* VOLUNTEER INCLUSION CRITERIA:

Volunteers will be able to enroll if they:

* Have the ability to understand and sign an informed consent.
* Are able and willing to give a blood sample.
* Are healthy as determined by study Investigator.
* Have no chronic diseases.
* Do not exhibit any clinical indications of diabetes.

PARTICIPANT INCLUSION CRITERIA:

Participants will be able to enroll if they:

* Have the ability to understand and sign an informed consent.
* Are able and willing to give a blood sample.
* Have a clinical diagnosis of diabetes based on any one of the following criteria:

  1. Documented history of plasma glucose value greater than or equal to 210 mg/dl on three different occasions.
  2. Fasting blood sugar greater than or equal to 150 mg/dl on three different occasions.
  3. Documented history of ketoacidosis.
  4. Insulin dependency.
  5. Documented history of abnormal glucose tolerance test.

EXCLUSION CRITERIA:

Neither volunteers nor participants will be eligible if they:

* Are under the age of 10.
* Have severe systemic disease(s) that compromise our ability to obtain an adequate examination.
* Have any of the following ocular characteristics or conditions in both eyes:

  1. Opacities of the ocular media, limitations or pupillary dilation or any other problems sufficient to preclude good, quality stereo fundus photographs.
  2. Ocular disease which confounds assessment of diabetic retinopathy such as advanced age-related macular degeneration, central serous choroidopathy, optic atrophy, retinal vein occlusion, active uveitis, significant explained or unexplained visual field loss, or any other type of retinopathy or retinal degeneration.
  3. Chronic requirement for any ocular medication for other diseases, such as glaucoma.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2000-05-23; Study Completion 2010-12-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Winocour PD. Platelet abnormalities in diabetes mellitus. Diabetes. 1992 Oct;41 Suppl 2:26-31. doi: 10.2337/diab.41.2.s26. PMID 1526332
- [Background] Lupu C, Calb M, Ionescu M, Lupu F. Enhanced prothrombin and intrinsic factor X activation on blood platelets from diabetic patients. Thromb Haemost. 1993 Oct 18;70(4):579-83. PMID 8115982
- [Background] Jaffe EA. Cell biology of endothelial cells. Hum Pathol. 1987 Mar;18(3):234-9. doi: 10.1016/s0046-8177(87)80005-9. PMID 3546072